CLINICAL TRIAL: NCT05650866
Title: Safety and Tolerability of a Novel Implantable Device for the Treatment of Erectile Dysfunction Following Radical Prostatectomy
Brief Title: Safety and Tolerability of a Novel Implantable Device for the Treatment of Erectile Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Comphya Australia (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-1.5400
Record Dates: First submitted 2022-11-28; First posted 2022-12-14 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Erectile Dysfunction Following Radical Prostatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Implanted group (Experimental): The study device will be implanted during the ongoing prostatectomy surgery. Participants will then be asked to activate it everyday.
  Interventions: Device: Activation of pro-erectile nerves within the pelvic plexus
- Control group (No Intervention): Participants in the control group will undergo standard prostatectomy and will not be implanted with the study device.

INTERVENTIONS:
Device: Activation of pro-erectile nerves within the pelvic plexus — The study device is an active implantable device. The device activates the cavernous nerves by delivering electrical pulses, to trigger an on-demand erection. The daily delivery of electrical pulses to the cavernous nerves will also allow participants to recover natural erectile function.
  Arms: Implanted group

SUMMARY:
The goal of this clinical trial is to assess if a new device is safe to use as a potential treatment for erectile dysfunction following radical prostatectomy.

The main questions it aims to answer are:

* Is the device safe?
* Does the device works well? Are the participants satisfied with the device?

Participants will be implanted with the device during the ongoing prostatectomy surgery and will be asked to complete the following tasks during 6 months follow-up:

* Come to the hospital for follow-up visits,
* Complete questionnaires,
* Activate the device every day,
* Measure erection hardness.

Researchers will compare an implanted group (participants having the device) with a control group (participants not having the device) to see if the device works well.

ELIGIBILITY:
Inclusion Criteria:

* Men of ages between 30-70 years;
* Men with indication for nerve-sparing prostatectomy surgery;
* Localised prostate cancer considered suitable for bilateral nerve sparing prostatectomy according to clinical criteria
* International Index of Erectile Function (IIEF-15) erectile function domain score equal to or greater than 26 prior prostatectomy;
* Men interested in minimizing the effect of radical prostatectomy on erectile function;
* Ability to read and understand patient information materials and willingness to sign a written informed consent.

Exclusion Criteria:

* Men with neurological disease, including a history of spinal cord injury or trauma;
* IIEF-15 erectile function domain score less than 26 prior prostatectomy;
* Failure to demonstrate adequate nocturnal erectile function prior prostatectomy;
* History of erectile dysfunction, priapism and Peyronie disease;
* History of previous pelvic surgery, trauma or irradiation therapy;
* Currently have an active implantable device;
* Patient diagnosed with neurologic degenerative diseases that may negatively impact erectile functions;
* Identification of technical or clinical limitation to properly apply the use of nerve-sparing techniques during operation;
* Inability to understand and demonstrate device use instructions;
* Patients with insulin-dependent diabetes who suffer peripheral neuropathy or other diabetes associated complications;
* Patient unwillingness to engage in sexual activity;
* Patient is currently participating in another clinical investigation that would serve as a contraindication to implant a neurostimulator device to augment erectile function;
* Have participated in any drug or device trial in the last 4 weeks or plan to participate in any other drug or device study during the next 24 months;
* Possess any other characteristics that, per the investigator's judgment, may increase the risk or impair data collection for the procedure/study;
* Patient is a member of a vulnerable population (Vulnerable participants include those who lack consent capacity, including the mentally ill, prisoners, cognitively impaired participants, and employee volunteers).

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender eligibility: male. Not based on self-representation of gender identity.
Enrollment: 20 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2025-05-19 (Estimated); Study Completion 2025-05-19 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events | 6 months
  Adverse events will be reported using MedDRA terminology.
Occurrence of surgical complications | 6 months
  Surgical complications will be ranked according to the Clavien-Dindo classification
Occurrence of device deficiencies | 6 months
  Device deficiencies will be systematically reported and recorded.
Pain | 6 months
  Patients will be asked to rate pain on a visual analog scale (from 0 to 10)

SECONDARY OUTCOMES:
Objective Device effectiveness | 6 months
  Erectile response obtained when activating the study device will be objectively assessed by measuring penile rigidity with the RigiScan device.
Subjective Device effectiveness | 6 months
  Erectile function will be subjectively assessed by asking participants to complete validated questionnaires (International Index of Erectile Function, IIEF-15 and Erection Hardness Score, EHS).
Erectile function recovery | 6 months
  Nocturnal penile erections will be assessed with the RigiScan device. Nocturnal erections reflect the extent of recovery of natural erectile function.
Delineation of the surgical implantation procedure | 6 months
  The surgeon will record information related to the implantation (duration, position of the device, grading ease of implantation steps, and any comments).

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - St. Vincent's Private Hospital, Fitzroy, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Australian Prostate Centre, North Melbourne, Victoria
  - Epworth HealthCare, Richmond, Victoria

IPD SHARING:
Plan to Share IPD: No